CLINICAL TRIAL: NCT03815578
Title: Evaluation of Pain Sensitization in Rheumatoid Arthritis: Analysis on a Cohort of Tofacitinib Treated Patients
Acronym: TOPRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2017/39
Record Dates: First submitted 2019-01-11; First posted 2019-01-24 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Rheumatoid Arthritis
Keywords: pain sensitization; Tofacitinib; miRNA
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Restraint, Physical; Blood Specimen Collection; Patient Reported Outcome Measures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rheumatoid Arthritis (RA) patients (Experimental): RA according to the ACR/EULAR 2010 classification criteria
  Interventions: Other: Clinical examination; Other: Pain assessment; Other: blood sample; Other: Patient Reported Outcomes

INTERVENTIONS:
Other: Clinical examination — * Number of painful joints,
  * Number of swollen joints,
  * Patient Global assessment VAS (0 - 100)
  * and Physician Global assessment VAS (0 - 100)
Other: Pain assessment — * Pressure Pain Thresholds (PPTs),
  * Mechanical Temporal Summation (MTS)
  * and Diffuse Noxious Inhibitory Control (DNIC)
Other: blood sample — 18 ml whole blood for ELISA analysis and miRNAs detection
Other: Patient Reported Outcomes — * Health Assessment Questionnaire (HAQ),
  * Rheumatoid Arthritis Impact of Disease score (RAID),
  * Daily joint pain intensity VAS (0-100),
  * Hospital Anxiety and Depression scale
  * and Coping Strategy Questionnaire.

SUMMARY:
Persistent pain and chronic fatigue are very common complaints in rheumatoid arthritis (RA) patients, whatever the anti-inflammatory treatment response. Interestingly, pain remaining despite good clinical response was associated with high disability and low inflammation at baseline, suggesting a mechanism of pain independent of inflammation in these patients. Such patients, with discordantly high patient-reported DAS28 components, fatigue and mood disturbance might represent a subgroup of RA patients who have specific clinical needs, not resolved by classical conventional or biologic DMARDs. In this way, neuropathic pain and pain sensitization have been demonstrated in 20 to 30% of RA patients, neuropathic pain scores being associated with worsen disease activity scores. Thus, pain sensitization may contribute to amplification of pain in active RA, and should be responsible for persisting pain and fatigue even after inflammation has resolved.

Pain sensitization is associated with neuroplastic changes in sensory pathways at peripheral and central levels. Interestingly, major mediators responsible for this neuroplasticity operate via a JAK/STAT signaling pathway, which is specifically targeted by new RA treatments. New drug targeting JAK/STAT signalling pathway have been recently designed for RA treatment, based on the implication of this pathway on the signaling of various cytokines implicated in the pathophysiology of RA, such as IL-6, IL-12, IL-23 and IFNs. Two Jak-inhibitors have been put on the market: Tofacitinib and Baricitinib. In randomized clinical trials, Tofacitinib have shown a remarkable efficacy on pain and other patient reported outcomes, suggesting a specific effect or jak-inhibitors on pain control. Recent data suggest that Jak-inhibitors could have a direct effect on sensory neurons.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 year-old ;
* Diagnosis of RA according to the ACR/EULAR 2010 classification criteria ;
* Active rheumatoid arthritis defined by a Disease Activity Score (DAS28) > 3.2 at inclusion ;
* Patient eligible for tofacitinib treatment in agreement with European treatment labelling and French recommendation for RA treatment ;
* Oral prednisone intake is allowed until 10 mg, stable for at least 1 week at study entry ;
* Starting tofacitinib treatment for an active RA defined by a DAS28-ESR > 3.2 ;
* Affiliated person or beneficiary of a social security scheme ;
* Having signed an informed consent (at the latest on the day of inclusion and before any examination required by research).

Exclusion Criteria:

* Diagnosis of a systemic autoimmune disease other than RA ;
* Peripheral neuropathy ;
* Centrally-acting pain medications use within 3 months of enrolment (amitriptyline, gabapentin, duloxetine), or during the study ;
* Any opioid use within 1 month of enrolment or during the study ;
* Corticosteroid treatment over 10 mg of prednisone or equivalent ;
* Patient who present contraindications to tofacitinib treatment ;
* Patient presenting with a history of active tuberculosis or chronic infectious disease with a need of regular use of antibiotic ;
* Patients with active bacterial or viral infection, or presenting with an episode of infection that required treatment with antibiotics within 30 days prior to screening ;
* Patient presenting with a history of lymphoma or leukaemia or other malignancy besides non-melanoma skin cancer within 5 years ;
* Patient presenting with any uncontrolled medical condition ;
* Pregnancy or breast-feeding ;
* Patient unable to understand and follow recommendations or unable to perform self-evaluation ;
* Patient who refuse to participate to the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2023-04-28 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Variation of the mean Pressure Pain Thresholds (PPTs) | At 6 months from baseline

SECONDARY OUTCOMES:
Variation of Mechanical Temporal Summation (MTS) | At 1, 3 and 6 months from baseline
Variation of Pressure Pain Thresholds (PPTs) | At 1, 3 and 6 months from baseline
Variation of Diffuse noxious inhibitory control (DNIC) values | At 1, 3 and 6 months from baseline
Variation of Daily joint pain intensity | At 1, 3 and 6 months from baseline
  daily evaluation of the previous 24h pain on a numeric pain scale 0 to 100
Disease activity evaluated by the Disease Activity Score on 28 joints (DAS28) | At 1, 3 and 6 months from baseline
  which take into account the number of painful joints (on 28 joints), the number of swollen joints (on 28 joints), the patient global assessment of disease activity (between 0 and 100), and the erythrocyte sedimentation rate.
Disease activity evaluated by the Simple Disease Activity Index (SDAI) | At 1, 3 and 6 months from baseline
  which take into account the number of painful joints (on 28 joints), the number of swollen joints (on 28 joints), the patient global assessment of disease activity (between 0 and 100), the physician global assessment of disease activity (between 0 and 100), and the C-reactive protein level.
Disease activity evaluated by the Clinical Disease Activity Index (SDAI) | At 1, 3 and 6 months from baseline
  which take into account the number of painful joints (on 28 joints), the number of swollen joints (on 28 joints), the patient global assessment of disease activity (between 0 and 100), and the physician global assessment of disease activity (between 0 and 100).
Health Assessment Questionnaire (HAQ) | At 1, 3 and 6 months from baseline
Rheumatoid Arthritis Impact of Disease score (RAID) | At 1, 3 and 6 months from baseline
Hospital Anxiety and Depression scale | At 1, 3 and 6 months from baseline
  HAD scale aims at evaluating anxiety and depression symptoms with two separate scores (between 0 and 21) estimated grace to 14 items (7 for anxiety and 7 for depression) ranged between 0 and 3
Coping Strategy Questionnaire: a 21-items self-report | At 1, 3 and 6 months from baseline
Levels of cytokines | At 3 and 6 months from baseline
Levels of neurotrophins | At 3 and 6 months from baseline
Levels of miR21, miR-124, miR-146a and miR-155 | At 3 and 6 months from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Thierry SCHAEVERBEKE, Prof, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - CHU de Bordeaux - Service de rhumatologie, Bordeaux
  - CHU de Limoges - service de rhumatologie, Limoges

IPD SHARING:
Plan to Share IPD: No